CLINICAL TRIAL: NCT05413668
Title: A Single Center, Double-Blinded, Phase 1a Randomized Study to Evaluate Safety and Pharmacokinetics of a New Manganese Based Magnetic Resonance Imaging (MRI) Contrast Agent, RVP-001, in Healthy Adult Subjects
Brief Title: First in Human Study of RVP-001, a New Manganese Based MRI Contrast Agent
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reveal Pharmaceuticals Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: RVL-101-22; R44CA268392 (NIH)
Record Dates: First submitted 2022-05-26; First posted 2022-06-10 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RVP-001 group (Experimental): 4 Cohorts of 6 subjects each will receive RVP-001 at doses of 2, 4, 7 and 12 mg Mn/kg.
  Interventions: Drug: RVP-001
- Placebo group (Placebo Comparator): 4 Cohorts of 2 subjects each will receive placebo (saline).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RVP-001 — Intravenous administration of RVP-001
  Other Names: MnPyC3A
  Arms: RVP-001 group
Drug: Placebo — Intravenous administration of saline placebo
  Other Names: saline
  Arms: Placebo group

SUMMARY:
The objectives of this trial are:

1. To evaluate the safety and tolerability of single ascending doses of RVP-001 in healthy adult volunteers
2. To determine the pharmacokinetics and elimination of RVP-001 in healthy adult volunteers.

DETAILED DESCRIPTION:
The first in human study is intended to evaluate the safety and tolerability of single ascending doses of RVP-001 in healthy adult volunteers, and to determine the pharmacokinetics and elimination of RVP-001 in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects
2. Healthy subjects aged 18 to 55 years inclusive
3. Suitable veins for phlebotomy, cannulation, or repeated venipuncture
4. Have a body mass index between 18 and 32 kg/m^2 (inclusive); weigh at least 55 kg.
5. Appropriately completed written informed consent prior to any study specific procedures.

Exclusion Criteria:

1. Any clinically significant abnormality or abnormal laboratory test results found during medical screening
2. Vital sign abnormalities at screening or admission
3. History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease; neurological or psychiatric disorder, as judged by the investigator
4. Positive pregnancy test at screening or admission
5. History of alcohol abuse
6. History of drug abuse
7. Use of nicotine-containing products within 12 months of study start
8. Use of medication except topical products without significant systemic absorption
9. Known allergies to any component of RVP-001
10. Subjects who have received any investigational product (IP) in a clinical research study within 5 IP half-lives or 30 days prior to first dose.
11. Donation of plasma within 7 days prior to dosing; significant donation or loss of blood within 30 days prior to the first dosing.
12. Any reason which, in the opinion of the Principal Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivasan Mukundan, MD, Study Director — Reveal Pharmaceuticals; Jeffrey Levy, MD, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- RVP-001: 2 mg Mn/kg: 6 subjects received RVP-001 in a single dose of 2 mg Mn/kg administered via automated injection pump.
- RVP-001: 4 mg Mn/kg: 6 subjects received RVP-001 in a single dose of 4 mg Mn/kg administered via automated injection pump.
- RVP-001: 7 mg Mn/kg: 6 subjects received RVP-001 in a single dose of 7 mg Mn/kg administered via automated injection pump.
- RVP-001: 12 mg Mn/kg: 6 subjects received RVP-001 in a single dose of 12 mg Mn/kg administered via automated injection pump.
- Placebo Group: Placebo
  Placebo: Intravenous administration of saline placebo
Period: Overall Study
Arm/Group | RVP-001: 2 mg Mn/kg | RVP-001: 4 mg Mn/kg | RVP-001: 7 mg Mn/kg | RVP-001: 12 mg Mn/kg | Placebo Group
Started | 6 | 6 | 6 | 6 | 8
Dosed | 6 | 6 | 6 | 6 | 8
Completed | 6 | 6 | 6 | 6 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Group: 8 subjects received placebo (saline) administered via automated injection pump
- Total: Total of all reporting groups
Arm/Group | RVP-001: 2 mg Mn/kg | RVP-001: 4 mg Mn/kg | RVP-001: 7 mg Mn/kg | RVP-001: 12 mg Mn/kg | Placebo Group | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 8 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 38.3 [22 to 55] | 35.3 [25 to 54] | 30.3 [22 to 35] | 44.3 [32 to 54] | 39.0 [30 to 52] | 38.53 [22 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 3 | 2 | 10
  Male | 5 | 4 | 4 | 3 | 6 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 6 | 6 | 8 | 32
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 3 | 0 | 3 | 7
  White | 5 | 6 | 3 | 6 | 5 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Body Weight [Mean (Full Range); unit: Kg] | 72.97 [62.8 to 96.3] | 77.57 [63.5 to 92.3] | 79.00 [58.8 to 92.8] | 76.83 [60.5 to 90.8] | 81.09 [67.7 to 90.5] | 77.72 [58.8 to 93.3]
Height [Mean (Full Range); unit: cm] | 167.5 [148 to 186] | 169.3 [160 to 180] | 170.8 [160 to 179] | 168.0 [156 to 182] | 171.0 [161 to 181] | 169.4 [148 to 186]
BMI [Mean (Full Range); unit: kg/m^2] | 26.03 [22.0 to 31.1] | 26.95 [23.0 to 30.4] | 26.93 [20.8 to 29.6] | 27.08 [24.9 to 29.3] | 27.66 [24.9 to 30.3] | 26.98 [20.8 to 31.1]

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter Cmax
Description: Cmax = maximum observed blood plasma concentration of RVP-001
Time Frame: pre-dose, 2, 5, 10, 20, 30 min and 1, 2, 4, 8, 12, 24, 48, 72, 96, 120 hours post-dose
Population: All subjects who received at least one dose of RVP-001 and had sufficient data to calculate at least one PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/mL
Groups:
- RVP-001: 7 mn Mn/kg: 6 subjects received RVP-001 in a single dose of 7 mg Mn/kg administered via automated injection pump.
Arm/Group | RVP-001: 2 mg Mn/kg | RVP-001: 4 mg Mn/kg | RVP-001: 7 mn Mn/kg | RVP-001: 12 mg Mn/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
nmol/mL | 264 (21.6) | 685 (31.1) | 992 (20.2) | 1960 (20.3)

2. Primary Outcome: PK Parameter Tmax
Description: tmax = time of maximum observed plasma concentration of RVP-001
Time Frame: pre-dose, 2, 5, 10, 20, 30 min and 1, 2, 4, 8, 12, 24, 48, 72, 96, 120 hours post-dose
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | RVP-001: 2 mg Mn/kg | RVP-001: 4 mg Mn/kg | RVP-001: 7 mn Mn/kg | RVP-001: 12 mg Mn/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours | 0.065 [0.04 to 0.09] | 0.085 [0.04 to 0.17] | 0.084 [0.03 to 0.17] | 0.091 [0.05 to 0.17]

3. Primary Outcome: PK Parameter t1/2
Description: t1/2 = terminal elimination half-life of RVP-001
Time Frame: pre-dose, 2, 5, 10, 20, 30 min and 1, 2, 4, 8, 12, 24, 48, 72, 96, 120 hours post-dose
Population: All subjects who received at least one dose of RVP-001 and had sufficient data to calculate at least one PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | RVP-001: 2 mg Mn/kg | RVP-001: 4 mg Mn/kg | RVP-001: 7 mn Mn/kg | RVP-001: 12 mg Mn/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours | 1.718 (7.4) | 1.765 (7.9) | 1.613 (7.0) | 1.839 (20.2)

4. Primary Outcome: PK Parameter Cl
Description: Cl = total body clearance calculated after a single IV administration of RVP-001
Time Frame: pre-dose, 2, 5, 10, 20, 30 min and 1, 2, 4, 8, 12, 24, 48, 72, 96, 120 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | RVP-001: 2 mg Mn/kg | RVP-001: 4 mg Mn/kg | RVP-001: 7 mn Mn/kg | RVP-001: 12 mg Mn/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mL/min | 122 (18.8) | 102 (6.4) | 122 (16.3) | 97.6 (13.3)

5. Primary Outcome: PK Parameter Vd
Description: Vd = volume of distribution calculated after a single IV administration of RVP-001
Time Frame: pre-dose, 2, 5, 10, 20, 30 min and 1, 2, 4, 8, 12, 24, 48, 72, 96, 120 hours post-dose
Population: All subjects who received at least one dose of RVP-001 and had sufficient data to calculate at least one PK parameter
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | RVP-001: 2 mg Mn/kg | RVP-001: 4 mg Mn/kg | RVP-001: 7 mn Mn/kg | RVP-001: 12 mg Mn/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Liters | 18.2 (17.8) | 15.6 (8.8) | 17.1 (18.4) | 15.5 (22.7)

6. Secondary Outcome: % RVP-001 Dose Excreted
Description: mean % of RVP-001 excreted from urine from 0 -120 hours post dose
Time Frame: pre-dose, 2, 5, 10, 20, 30 min and 1, 2, 4, 8, 12, 24, 48, 72, 96, 120 hours post-dose
Measure: Mean (Standard Deviation); unit: Mean % of dose recovered 0-120 hrs
Arm/Group | RVP-001: 2 mg Mn/kg | RVP-001: 4 mg Mn/kg | RVP-001: 7 mn Mn/kg | RVP-001: 12 mg Mn/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Mean % of dose recovered 0-120 hrs | 66.398 (7.372) | 73.623 (7.768) | 80.924 (12.347) | 74.90 (15.230)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from signing of consent to last study visit - approximately 7 days.
Description: Adverse events were defined as "Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research."
Groups:
- Placebo Group: 8 subjects received placebo (saline) via automated injection pump
Arm/Group | RVP-001: 2 mg Mn/kg | RVP-001: 4 mg Mn/kg | RVP-001: 7 mg Mn/kg | RVP-001: 12 mg Mn/kg | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 1/6 | 2/6 | 2/6 | 0/6 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RVP-001: 2 mg Mn/kg (N=6) | RVP-001: 4 mg Mn/kg (N=6) | RVP-001: 7 mg Mn/kg (N=6) | RVP-001: 12 mg Mn/kg (N=6) | Placebo Group (N=8)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT05413668/Prot_SAP_000.pdf